CLINICAL TRIAL: NCT04514718
Title: Short- and Medium-term Safety/Effectiveness Analysis of Low Energy Holmium Laser Enucleation of the Prostate (HoLEP)
Brief Title: Low Energy HoLEP on IPSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Seung-June Oh, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-2002-054-1100
Record Dates: First submitted 2020-08-13; First posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Prostate Hyperplasia; Prostatic Hypertrophy; Surgery; Bladder Outlet Obstruction; Quality of Life; Complication of Surgical Procedure
MeSH Terms: conditions — Prostatic Hyperplasia; Urinary Bladder Neck Obstruction | interventions — Lasers, Solid-State

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low energy holmium laser (Active Comparator): 30 watts
  Interventions: Device: Holmium laser
- high energy holmium laser (Active Comparator): 80-100 watts
  Interventions: Device: Holmium laser

INTERVENTIONS:
Device: Holmium laser — low energy holmium laser

SUMMARY:
The purpose of this study is to prove that low-energy (30W) Holmium laser prostatectomy (Holeb) is not inferior to high-energy (100W) Holmium laser prostatectomy (safety and effectiveness)

DETAILED DESCRIPTION:
1. Overview of the study Research design: prospective, single-arm blind randomized control study, non-inferiority study Study Period: 12 months since IRB approval date Subject: Patients with benign prostatic hyperplasia Number of study subjects: 90 Vulnerable Subjects: None
2. Background and purpose of the study

1) Research background

1. Overview and main symptoms of prostatic hyperplasia (BPH)

   -The prostate is a male reproductive organ located in the lower bladder. Benign prostatic hyperplasia (BPH) causes lower urinary tract symptoms (LUTS) due to bladder outlet obstruction.
   * The prevalence of prostatic hyperplasia is known to reach 37% in the 50s, 49% in the 60s, and 70% in the 70s; a disease with a very high incidence in long-aged men.
   * BPH is a disease directly related to the quality of life that interferes with the patient's social life, sexual life, and daily life. If it persists for a long time, it may cause bladder stones, hematuria, and even renal dysfunction, so timely treatment is absolutely necessary.
2. Surgical Treatment of BPH

   -Surgical treatment is recommended for an enlarged prostate that is not treated with drugs, and transurethral surgery using an endoscope is recommended for standard surgery for an enlarged prostate.
   * Transurethral surgery for BPH varies from traditional transurethral resection of the prostate (TURP) to holmium laser enucleation of the prostate (HoLEP).
   * HoLEP has a sharp increase in the number of surgeries worldwide due to its low recurrence rate, high efficiency, and high patient satisfaction;
   * Since its first introduction in 2008 in Korea, the number and rate of surgeries have been steadily increasing. The total number of surgery for BPH is equivalent to about 10,000 cases per year. TUR-P and KTP laser surgery are on a decreasing trend, while HoLEP is on an increasing trend.
3. The importance of HoLEP

   -HoLEP is a surgery to completely remove prostate tumors using a Holmium-YAG Laser of 2100nm wavelength.

   -The tissue penetration depth of the Holmium laser is less than 0.44mm, enabling sharp incisions, and has the advantage of less bleeding than traditional transurethral prostatectomy.

   -The surgery principle of HoLEP is fundamentally different from TUR-P and KTP laser prostate vaporization. TUR-P and KTP laser prostatectomy aim to remove part of the prostate tumor, whereas HoLEP performs complete removal of the prostate tumor according to the anatomical structure.

   -HoLEP consists of two steps, and the first step consists of an enucleation step in which the prostate tumor is completely removed and placed in the bladder, and a morcellation step in which the enucleated adenoma tissue is morcellated and removed.
   * HoLEP is relatively safe compared to other transurethral surgery and can completely remove prostate adenoma, so it has a low recurrence rate and the patient's satisfaction with surgery is over 90%, making it the next-generation standard treatment for BPH.
4. Low energy HoLEP related research and clinical status -HoLEP is mainly applied to treatment with 80-100 Watt high energy equipment. High-energy HoLEP has the advantage of removing prostate tumors in a short time, but there are problems of frequent laser fiber damage, device shutdown problems, and possible bladder damage due to scattered lasers.

   * In 2008, Rassweiller et al. proposed the possibility of clinical application of low energy HoLEP by applying a 40 Watt Holmium laser. Since then, prospective studies have been published sporadically. In 2018, a prospective randomized study that compared and analyzed the prostate removal efficiency of 50 Watt laser and 100 Watt laser in a total of 121 patients was the latest and largest study and confirmed that low-energy prostatectomy is not inferior to the high-energy procedure. And proved its clinical safety.
   * In theory, low-energy HoLEP reduces dysuria immediately after surgery and storage symptoms after surgery. It is estimated to be advantageous in preserving erectile function.
   * The research team is the first in the world to compare the safety and usefulness of 30 Watt HoLEP with 100 Watt HoLEP through prospective, non-inferiority studies.

     2) Research goal The final purpose of the study: To prove that the low-energy (30Watt) HoLEP is not inferior to the high-energy (100Watt) HoLEP in short-term and mid-term surgical results (safety and effectiveness).

Detailed research objectives:

1. Compare short-term (2 weeks-1 months) surgical outcomes/surgical complications of low energy HoLEP with high energy HoLEP.
2. Compare the mid-term (3, 6 months) surgical outcomes/surgical complications of low-energy HoLEP with high-energy HoLEP.

3) Selection criteria, exclusion criteria, the target number of subjects and basis for calculation

* Selection criteria Men over 50 Patients receiving HoLEP due to an enlarged prostate Patients who fully understood and agreed to the study
* Exclusion criteria Patients with neuropathy that may adversely affect the urination function (Parkinson's disease, dementia, etc.) Patients with acute urinary retention within the last month Patients with symptomatic urinary tract infection In case there are other factors that can significantly affect treatment results at the discretion of the researcher

  (2) Number of research subjects About 90 patients
* The basis for calculating the number of subjects This study aims to prospectively enroll and randomize prostatectomy patients, and then compare the results of the treatment at 6 months after the maximum operation to confirm non-inferiority.

The current standard is a method using a high-energy holmium laser, and the treatment results for 6 months after surgery have been published through many studies. The research team wants to confirm the surgical outcome as a decrease in the International Prostate Symptom Score (IPSS). After 6 months of predicted high-energy HoLEP, IPSS in other literature (5.1 ± 5.0), 6 months after the expected of low-energy HoLEP. IPSS is estimated from the most recently published academic paper (5.0 ± 5.0).

Alpha (0.15) and Beta (0.8) were calculated, and the non-inferior margin was set to 3. The estimated number of subjects is calculated by considering the 20% drop-out rate. Statistics for calculating the number of subjects are calculated using PASS 2019.

Considering drop-out 20%, it is necessary to recruit 25-114 patients (total 50-114) per group to conduct the study.

This organization is an organization that implements about 20-30 HoLEP cases per month, and a follow-up period of up to 6 months is required to announce short-term and mid-term results. Therefore, the actual patient enroll period is estimated to be up to 6 months. It is expected that 120-180 patients can undergo surgery during the recruitment period of up to 6 months, and assuming that only 60% of patients will participate in the study based on the median of about 150, a total of 90 patients, about 45 for each group. It is judged realistic to conduct a study with 3 patients.

4. Research method

1. Specific research method Since the researchers have already published dozens of studies related to HoLEP surgery, we are securing a systematic preoperative examination/postoperative follow-up process. The preoperative examination/postoperative follow-up protocol of high energy HoLEP surgery, which was previously performed, will be used as it is, but the study will be conducted by adding only the preoperative randomization process.

   -Pre-screening: After making operation in the outpatient clinic, before hospitalization, it is checked whether it is subject to enroll according to the patient record.

   -Random allocation: Using R package (RandomizeR), low energy HoLEP, and high energy HoLEP is randomly assigned.

   -Pre-Op work-up & Operation: This item is irrelevant to Randomization and is a situation where you do not know who will undergo surgery, so it is considered a normal treatment process and proceeds according to the existing process.
   * Monitoring: It is planned to perform research ethics, safety, and monitoring work independently from the researcher by requesting the Medical Device Innovation Center.
   * Clinical trial insurance: In case of adverse side effects to patients, the company plans to subscribe to clinical trial liability insurance through the Medical Device Innovation Center to notify the patient of the procedures and details of the clinical trial damage relief.
   * Compensation: There is no monetary incentive for research participants, and the research team will pay 30,000 won of transportation and inspection costs (160,000 won) per visit during the participation period of visit #1-#3.
2. Test drug administration/dosage, administration/use method, combination therapy, reasons for selection when using a reference drug None
3. Observation items, clinical test items and observation test methods Primary endpoint: 3-6 month questionnaire (International Prostate Symptom Score, IPSS) total score

Secondary endpoint:

1) Surgery day: surgery time, total energy, resected prostate volume, immediate complication

1) 2 weeks after surgery: questionnaire (IPSS-subscore, IPSS-QoL, OABSS total score), Qmax, 2) post voided residual urine volume, Clavian-Dindo complication classification 3) 3, 6 months after surgery: questionnaire (IPSS-total, IPSS subscore, IPSS-QoL, OABSS total score), Qmax, post voided residual urine volume, Clavian-Dindo complication classification, urine test (urinalysis, urine microscopy), serum PSA level

4) Effect evaluation criteria, evaluation method Efficacy

1. Statistical analysis of low-power HoLEP is not inferior in short-term (2wk/1month) and mid-term (3-6 months) IPSS.
2. Uroflowmetry (UFM) and non-inferiority of post voided residual (PVR) were verified in urinalysis.
3. 3 months/6 months U/A, micro, 6 months PSA
4. Non-inferiority was verified in terms of improving the patient's QoL.
5. To verify the non-inferiority of the storage symptom subscore after the patient's surgery.

Safety:

1. The safety of HoLEP has been revealed to some extent through overseas research results, so animal testing is not required. For the safety, all safety issues that occurred using the Clavian-Dindo grade, which are commonly used clinically in human studies, were recorded and compared and analyzed.
2. If adverse events that occurred immediately after surgery and during up to 3 visits were recorded and there was a statistically significant difference in complications of Grade III-IV, it was judged that there was a safety problem.

4) The difference between existing treatment and research Existing studies comparing low energy HoLEP surgery and high energy HoLEP are mostly retrospective studies, and two prospective studies have been performed.

One of the two prospective studies involved 54 patients and had no active control group.

The most recent study was RCT with 121 subjects, but it was a study comparing 50W laser and 100W laser.

This study is the first in the world to compare 30W laser and 100W laser, and it is a prospective, RCT that recruits 90 patients, and it is judged that the results of the study can provide important medical evidence for the safety and effectiveness of low-energy HoLEP surgery.

ELIGIBILITY:
* Selection criteria Men over 50 Patients receiving HoLEP due to an enlarged prostate Patients who fully understood and agreed to the study
* Exclusion criteria Patients with neuropathy that may adversely affect the urination function (Parkinson's disease, dementia, etc.) Patients with acute urinary lung disease within the last month Patients with symptomatic urinary tract infection In case there are other factors that can significantly affect treatment results at the discretion of the researcher

Ages: 50 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-08-24 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
IPSS total score | baseline, postoperative 3 months, and 6 months
  International Prostate Symptom Score

SECONDARY OUTCOMES:
surgery time, total energy, resected prostate volume, immediate complication | Surgery day
  surgery related outcomes
IPSS-subscore, IPSS-QoL, OABSS total score | baseline, postoperative 3 months, and 6 months
  International Prostate Symptom Score
Qmax, post voided residual urine volume | baseline, postoperative 3 months, and 6 months
  efficacy outcomes

IPD SHARING:
Plan to Share IPD: No